CLINICAL TRIAL: NCT05088785
Title: Dynamic and Test-retest Whole Body [18F]FES PET Imaging in Patients With Metastatic ER+ Breast Cancer
Acronym: FEStastic
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, C. Menke- van der Houven van Oordt, Principal investigator, Amsterdam UMC, location VUmc
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: NL76658.029.21
Record Dates: First submitted 2021-10-07; First posted 2021-10-22 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part A: dynamic FES PET imaging (Experimental): All patients included in part A will receive a dynamic FES PET/CT scan.
  Interventions: Drug: FES
- Part B: whole body static FES PET imaging (Experimental): All patients included in part B will receive a whole body static FES PET/CT scan twice within 1 week.
  Interventions: Drug: FES

INTERVENTIONS:
Drug: FES — [18F]FES PET imaging.

SUMMARY:
16a-18F-fluoro-17b-estradiol ([18F]FES) is radioactive labeled estradiol, developed for in vivo visualization of the estrogen receptor (ER) using positron emission tomography (PET). To date, [18F]FES PET has been mainly explored as a diagnostic imaging tool to assess ER expression, thereby identifying locations of disease and their potential sensitivity to endocrine therapy, respectively. The primary aim of this project is to extend the application of [18F]FES PET as a baseline diagnostic imaging biomarker for ER expression to use it as an (early) treatment response marker. However, for such an application, visual assessment alone may not be sufficient and a more rigorous quantitative image analysis is needed. Therefore, in this project we shall first derive the optimal pharmacokinetic model for full quantitative analysis of [18F]FES uptake and, subsequently, we shall assess the validity of simplified, clinically feasible, quantitative parameters of [18F]FES uptake in 5 patients with metastatic estrogen receptor positive (ER+) breast cancer (part A). In addition, the repeatability of these simplified parameters will then be investigated in another 10 patients (part B).

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven metastatic ER+ (>10% positive stained cells using immunohistochemistry) breast cancer on the latest biopsy
* Postmenopausal females aged 18 years or older at screening. Postmenopausal status is defined as one of the following:

  1. age ≥60 years
  2. age <60 years and amenorrhea for >12 months in the absence of interfering hormonal therapies (such as LH-RH agonists and ER-antagonists)
  3. patient age <60 years using LH-RH agonists should continue LH- RH-agonists until after the PET procedures
  4. previous bilateral oophorectomy or medically confirmed ovarian failure
* [18F]FDG PET, CT and/or a bone scan should be performed as part of routine clinical staging (≤4 weeks prior to screening)
* Patients should have metastases in the scanning field of view, all located outside of the liver
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0-2
* Estimated glomerular filtration rate (eGFR) ≥30 ml/min
* Written and signed informed consent

Exclusion Criteria:

* History with another cancer within the last 5 years, except cancer treated with curative intent and no evidence of disease as judged by the treating physician
* Use of selective estrogen receptor modulators (SERMs) or downregulators (SERDs) for current breast cancer such as Tamoxifen/Fulvestrant (≤5 weeks prior to screening) or investigational drug therapy
* Pregnancy or lactating women
* Any medical, psychological or social condition that may interfere with the subject's safety and participation in the study, will lead to exclusion from this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females only.
Enrollment: 15 (Estimated)
Dates: Start 2021-10-11 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
FES uptake in lesions: Ki (net influx rate) or VT (volume of distribution) values | 1 year
  FES uptake in lesions will be expressed as Ki or VT values

SECONDARY OUTCOMES:
SUV and TBR values | 1 year.
  Quantification of FES uptake in lesions will be assessed by determining standardized uptake values and tumor-to-blood ratios.

OTHER OUTCOMES:
SUV and TBR values | 1 year.
  Repeatability of standardized uptake values and tumor-to-blood ratios will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC - location VUmc, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No